CLINICAL TRIAL: NCT05895630
Title: Interactive and Adapted Physical Exercise for the Remote Management of Chronic Low Back Pain
Brief Title: Online Physical Exercise for Chronic Low Back Pain
Acronym: CLBPEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathieu Roy (Other)
Collaborators: Université de Montréal (Other); Université du Québec a Montréal (Other); Concordia University, Montreal (Other); Université du Québec à Trois-Rivières (Other); Institut Universitaire de Gériatrie de Montréal (Other)
Responsible Party: Sponsor-Investigator, Mathieu Roy, Assistant Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLBPEO
Record Dates: First submitted 2023-05-03; First posted 2023-06-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low-back Pain
Keywords: Physical exercise; Telehealth; Remote interventions; Motivation; Proof-of-concept
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Three-arm parallel randomized controlled trial
Who Masked: Participant
Masking Description: Participants will not be informed about the comparison arms, or about the specific aims of the study at comparing outcomes from two different types of online interventions. They will also not be made aware of the fact that the waitlist group will be compared to the intervention groups. However, it is not possible to mask completely participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive (Experimental): The sessions will be given in groups of 5 to 10 people and will be interactive via Zoom (link will be sent to them by email). They will last 1h30min and will consist of 60min of physical activity, preceded and followed by 15 optional minutes of virtual social interaction with the kinesiologist and the other members of the group. Finally, if the participants are unable to attend the group session, a video of the course given will be available for them to follow afterwards via a website.
  Interventions: Behavioral: Interactive physical exercise
- Video (Experimental): The sessions will be done individually without interaction via pre-recorded videos. The videos demonstrate specific classes provided to the patients in this arm by a kinesiologist. Participants will be able to contact the kinesiologist by phone or email to ask questions about the sessions. The sessions will last 1h30min.
  Interventions: Behavioral: Video physical exercise
- Control (No Intervention): The control will be instructed to continue their lifestyle habits throughout the study. These participants will not receive any intervention until their outcome measures at baseline and follow-up are recorded. At this point their participation is completed and they will be offered one of the two physical exercise programs. Therefore, this arm will be acting like a waitlist group.

INTERVENTIONS:
Behavioral: Interactive physical exercise — Interactive remote sessions of physical exercise in groups of 10 patients. The sessions are categorized by level 1, 2 or 3 and the allocation to this level is decided according to a decision tree taking into account the mobility profile (balance and cardiomuscular health). The intervention will last 12 weeks. The sessions will be delivered 3 times per week (Monday, Wednesday, Friday) offering a total of approximately 180 min/week.
  Arms: Interactive
Behavioral: Video physical exercise — Individual remote sessions of physical exercise based on pre-recorded videos. The video sessions are categorized by level 1, 2 or 3 and the allocation to this level is decided according to a decision tree taking into account the mobility profile (balance and cardiomuscular health). The videos will be delivered 3 times per week (Monday, Wednesday, Friday) offering a total of approximately 180 min/week.
  Arms: Video

SUMMARY:
This study aims to evaluate the effects of technology-based interventions, specifically web-based platforms, on outcomes of patients with chronic low back pain. The objectives are to develop and evaluate the feasibility and effectiveness of these interventions, and to examine factors such as age and gender on implementation and adherence. It consists of an interventional proof-of-concept pilot study with 45 participants randomly divided into 3 groups: an interactive physical activity group, a pre-recorded video physical activity group, and a control group. Assessments will be conducted at weeks 0 and 12 to measure pain intensity with the Canadian adaptation of the National Institutes of Health minimal dataset for chronic low back pain.

DETAILED DESCRIPTION:
Technology-based interventions, specifically web-based platforms, have been used during the pandemic and, to a lower extent, prior to it, to maintain and improve physical and mental health while avoiding physical contact and therefore, risk of contagion, but also facilitating access to services such as psychotherapy or rehabilitation. Specifically, remote interventions have shown to be effective in the management of symptoms of people with chronic musculoskeletal pain, including chronic low back pain (CLBP). The objectives are to develop and evaluate the feasibility and effectiveness of these interventions, and to examine factors such as age and gender on implementation and adherence, as well as to validate the effectiveness of the interventions in improving CLBP outcomes and compare the effects of two different modalities of remote intervention (interactive and pre-recorded videos) against a waitlist control group.

The study is an interventional proof-of-concept pilot study. Participants will be 45 people with CLBP aged 18 to 80 years who are able to consent, have no contraindication to physical activity, and can communicate, read, and understand French. Participants will be randomly divided into 3 groups: an interactive physical activity group, a video physical activity group, and a control group. Recruitment will be done from participant pools of the Quebec Pain Research Network, the Centre de Recherche de l'Institut Universitaire de Gériatrie de Montréal (CRIUGM), the Association Québécoise de la Douleur Chronique, and former participants of the laboratory's research projects. The intervention will last 12 weeks and consist of 3 physical activity sessions per week for the intervention groups. The interactive group sessions will be live via Zoom and the video sessions will consist of be pre-recorded videos. The control group will be instructed to continue their lifestyle habits throughout the study.

Assessments will be conducted at weeks 0 and 12 via videoconference, telephone or lime-survey format to measure physical health, mental health, lifestyle, and quality of life. It will also evaluate the feasibility and adherence of the interactive or video technology. The study will also take into account age, gender and baseline pain intensity as potential confounding factors, by introducing them as covariates. We will use ANOVAs to compare the effects of the intervention on the variables of interest between groups. The primary variable will be pain intensity from the National Institutes of Health minimum dataset for chronic low back pain. Other variables form this dataset will be explored as secondary outcomes, along with variables related to physical performance. The study aims to recruit 60 participants, with a 25% dropout rate, to have a sample size of 45 participants completing the project in order to detect a small effect size.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low back pain, lasting for more than 6 months
* To have an internet connection and access to a computer with webcam or tablet
* To be able to follow a physical activity program

Exclusion Criteria:

* Being under 18 years of age or over 80 years of age
* A history of psychiatric or neurological illness
* Presentation of neuropathic signs (radiating pain that spreads to the knee and leg (http://www.physio-pedia.com/Red_Flags_in_Spinal_Conditions)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline low back pain intensity at 12 weeks | Baseline and 12 weeks
  Pain intensity perceived on average for the previous 7 days, reported in an 11-point numerical rating scale from 0 (no pain) to 10 (maximum imaginable pain).

SECONDARY OUTCOMES:
Change from baseline pain spread at 12 weeks | Baseline and 12 weeks
  Has back pain spread down the leg(s) during the past 2 weeks, Yes/No/Not sure. Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline stomach pain at 12 weeks | Baseline and 12 weeks
  How much stomach pain bothered the patient during the past 4 weeks (Not bothered at all/Bothered a little/Bothered a lot). Item from the NIH (National Institutes of Health) Minimum Dataset for chronic low back pain
Change from baseline non-spine pain at 12 weeks | Baseline and 12 weeks
  How much pain in the arms, legs, or joints other than the spine of back bothered the patient during the past 4 weeks (Not bothered at all/Bothered a little/Bothered a lot). Item from the NIH (National Institutes of Health) Minimum Dataset for chronic low back pain
Change from baseline headache at 12 weeks | Baseline and 12 weeks
  How much headaches have bothered the patient during the past 4 weeks (Not bothered at all/Bothered a little/Bothered a lot). Item from the NIH (National Institutes of Health) Minimum Dataset for chronic low back pain
Change from baseline widespread pain at 12 weeks | Baseline and 12 weeks
  How much widespread pain (pain all over the body) has bothered the patient during the past 4 weeks (Not bothered at all/Bothered a little/Bothered a lot). Item from the NIH (National Institutes of Health) Minimum Dataset for chronic low back pain
Change from baseline opioid use at 12 weeks | Baseline and 12 weeks
  Has the patient used opioids (Yes/No/Not sure). Medical interventions item from the NIH Minimum Dataset for chronic low back pain
Change from baseline injection use at 12 weeks | Baseline and 12 weeks
  Has the patient used injections (epidural, facet) (Yes/No/Not sure). Medical interventions item from the NIH Minimum Dataset for chronic low back pain
Medical interventions: exercise therapy | Baseline
  Has the patient used exercise therapy (Yes/No/Not sure). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline psychological counseling use at 12 weeks | Baseline and 12 weeks
  Has the patient used psychological counseling such as cognitive behavioral therapy (Yes/No/Not sure). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline pain interference with day-to-day activities at 12 weeks | Baseline and 12 weeks
  Interference perceived on average for the previous 7 days, reported in an 5-point numerical rating scale from 1 (no interference) to 5 (maximum imaginable interference). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline pain interference with work around home at 12 weeks | Baseline and 12 weeks
  Interference perceived on average for the previous 7 days, reported in an 5-point numerical rating scale from 1 (no interference) to 5 (maximum imaginable interference). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline pain interference with ability to participate in social activities at 12 weeks | Baseline and 12 weeks
  Interference perceived on average for the previous 7 days, reported in an 5-point numerical rating scale from 1 (no interference) to 5 (maximum imaginable interference). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline pain interference with household chores at 12 weeks | Baseline and 12 weeks
  Interference perceived on average for the previous 7 days, reported in an 5-point numerical rating scale from 1 (no pain) to 5 (maximum imaginable interference). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline physical function (household chores) at 12 weeks | Baseline and 12 weeks
  Current ability to perform household chores, reported in an 5-point Likert scale (Without any difficulty, With a little difficulty, With some difficulty, With much difficulty, Unable to do). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline physical function (ability to go up and downstairs) at 12 weeks | Baseline and 12 weeks
  Current ability to go up and downstairs, reported in an 5-point Likert scale (Without any difficulty, With a little difficulty, With some difficulty, With much difficulty, Unable to do). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline physical function (ability to go for a walk for at least 15 minutes) at 12 weeks | Baseline and 12 weeks
  Current ability to go for a walk for at least 15 minutes, reported in an 5-point Likert scale (Without any difficulty, With a little difficulty, With some difficulty, With much difficulty, Unable to do). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline physical function (ability to run errands and shop) at 12 weeks | Baseline and 12 weeks
  Current ability to run errands and shop, reported in an 5-point Likert scale (Without any difficulty, With a little difficulty, With some difficulty, With much difficulty, Unable to do). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline feelings of depression (worthlessness) at 12 weeks | Baseline and 12 weeks
  Feeling worthless in the past 7 days, reported in an 5-point Likert scale (Never, Rarely, Sometimes, Often, Always). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline feelings of depression (helplessness) at 12 weeks | Baseline and 12 weeks
  Feeling helpless in the past 7 days, reported in an 5-point Likert scale (Never, Rarely, Sometimes, Often, Always). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline feelings of depression at 12 weeks | Baseline and 12 weeks
  Feeling depressed in the past 7 days, reported in an 5-point Likert scale (Never, Rarely, Sometimes, Often, Always). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline feelings of depression (hopelessness) at 12 weeks | Baseline and 12 weeks
  Feeling hopeless in the past 7 days, reported in an 5-point Likert scale (Never, Rarely, Sometimes, Often, Always). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline sleep quality at 12 weeks | Baseline and 12 weeks
  Sleep quality in the past 7 days, reported in an 5-point Likert scale (Very poor, Poor, Fair, Good, Very good). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline quantity of refreshing sleep at 12 weeks | Baseline and 12 weeks
  Refreshing sleep in the past 7 days, reported in an 5-point Likert scale (Not at all, A little bit, Somewhat, Quite a bit, Very much). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline extent of problems with sleep at 12 weeks | Baseline and 12 weeks
  Problem with sleep in the past 7 days, reported in an 5-point Likert scale (Not at all, A little bit, Somewhat, Quite a bit, Very much). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline difficulty falling asleep at 12 weeks | Baseline and 12 weeks
  Difficulty falling asleep in the past 7 days, reported in an 5-point Likert scale (Not at all, A little bit, Somewhat, Quite a bit, Very much). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline absenteeism and compensation benefits (time off work) at 12 weeks | Baseline and 12 weeks
  I have been off work or unemployed for 1 month or more due to low back pain (Yes/No/NA). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline absenteeism and compensation benefits (disability/compensation) at 12 weeks | Baseline and 12 weeks
  I receive or have applied for disability or workers compensation benefits because I am unable to work due to low back pain (Yes/No/NA). Item from the NIH Minimum Dataset for chronic low back pain
Baseline low back pain-related lawsuits and legal claims | Baseline
  Are you involved in a lawsuit or legal claim related to your low back problem? (Yes/No/NA). Item from the NIH Minimum Dataset for chronic low back pain
Follow-up low back pain-related lawsuits and legal claims | 12 weeks
  Are you involved in a lawsuit or legal claim related to your low back problem? (Yes/No/NA). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline kinesiophobia at 12 weeks | Baseline and 12 weeks
  Its not really safe for a person with my low back problem to be physically active (Agree/Disagree). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline catastrophizing at 12 weeks | Baseline and 12 weeks
  I feel that my low back pain is terrible and never going to get any better (Agree/Disagree). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline substance abuse (item 1) at 12 weeks | Baseline and 12 weeks
  Have you consumed alcohol or used drugs more than you meant to? (Never/Rarely/Sometimes/Often). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline substance abuse (item 2) at 12 weeks | Baseline and 12 weeks
  Have you felt you wanted or needed to cut down on your drinking or drug abuse? (Never/Rarely/Sometimes/Often). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline cigarette smoking at 12 weeks | Baseline and 12 weeks
  How would you describe your cigarette smoking? (Never smoked/Current smoker/Used to smoke, but have now quit). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline Body Mass Index group at 12 weeks | Baseline and 12 weeks
  Body Mass Index Group (Normal weight/Underweight/Overweight/Obesity I/Obesity II/Obesity III). Item from the NIH Minimum Dataset for chronic low back pain
Change from baseline Short Physical Performance Battery (SPPB) test score at 12 weeks | Baseline and 12 weeks
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. The scores range from 0 (worst performance) to 12 (best performance). Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Timed Up and Go (TUG) test score at 12 weeks | Baseline and 12 weeks
  TUG test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. Measured in seconds. Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Unipedal Stance test score at 12 weeks | Baseline and 12 weeks
  Unipedal stance test. Functional test where subjects are required to stand on one leg with eyes open, and if possible with eyes closed. It is timed in seconds. Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Lower Limb Strength test score at 12 weeks | Baseline and 12 weeks
  The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds (measured in absolute number of repetitions). Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Lower Limb Strength Takai test score at 12 weeks | Baseline and 12 weeks
  The Takai test is a 10 repetition chair stand, which involves recording the time it takes a person to complete 10 sit-to-stand repetitions (measured in seconds). Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Gait Speed test score at 12 weeks | Baseline and 12 weeks
  Consists on walking 4 meters at the fastest speed possible, measured in seconds. Patients are also requested to rate the intensity of their low back pain before and after performing this test, in an 11-point numeric rating scale from 0 (no pain) to 10 (maximum imaginable pain).
Change from baseline Rapid Assessment of Physical Activity (RAPA) test score at 12 weeks | Baseline and 12 weeks
  RAPA scale uses 7 items rated from 1 to 7 points, with the respondent's score categorized into one of five levels of physical activity: 1 = sedentary, 2 = underactive, 3 = regular underactive (light activities), 4 = regular underactive, and 5 = regular active.
Change from baseline International Physical Activity Questionnaire (IPAQ) test score at 12 weeks | Baseline and 12 weeks
  The International Physical Activity Questionnaire is a 27-item self-reported measure of physical activity. It measures duration (minutes) and frequency (days) of physical activity in the last 7 days in domains of: Job-related, Transportation, Housework, house maintenance, caring for family, Recreation, sport, and leisure-time, Time spent sitting. The scoring provides a result in metabolic equivalent minutes a week

OTHER OUTCOMES:
Pain intensity before each training session | Assessed before each of the 36 training sessions
  Participants will be asked to rate in an 11-point numerical rating scale from 0 (no pain) to 10 (maximum imaginable pain), the low back pain intensity perceived while standing, lying down and walking, before and after each training session
Pain intensity after each session | Assessed after each of the 36 training sessions
  Participants will be asked to rate in an 11-point numerical rating scale from 0 (no pain) to 10 (maximum imaginable pain), the low back pain intensity perceived while standing, lying down and walking, before and after each training session
Pain intensity during the performance of physical tests at baseline | Baseline
  Participants will be asked to rate in an 11-point numerical rating scale from 0 (no pain) to 10 (maximum imaginable pain), the low back pain intensity perceived during the SPPB, TUG, balance, lower limb strength and gait speed tests.
Pain intensity during the performance of physical tests at follow-up | 12 weeks
  Participants will be asked to rate in an 11-point numerical rating scale from 0 (no pain) to 10 (maximum imaginable pain), the low back pain intensity perceived during the SPPB, TUG, balance, lower limb strength and gait speed tests.
Program adherence | 12 weeks
  Adherence to the exercise programs will be assessed using the percentage of sessions attended. Participation ≥ 75% is considered necessary to be able to deem the program complete. In addition, a minimum of 66% of adherence (4/6 sessions) during the last two weeks will be required.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Roy, PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - McGill University, Montreal, Quebec
  - Centre de recherche de l'Institut universitaire de gériatrie de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips K, Clauw DJ. Central pain mechanisms in chronic pain states--maybe it is all in their head. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):141-54. doi: 10.1016/j.berh.2011.02.005. PMID 22094191
- [Background] Lauze M, Martel DD, Aubertin-Leheudre M. Feasibility and Effects of a Physical Activity Program Using Gerontechnology in Assisted Living Communities for Older Adults. J Am Med Dir Assoc. 2017 Dec 1;18(12):1069-1075. doi: 10.1016/j.jamda.2017.06.030. Epub 2017 Aug 14. PMID 28818422
- [Background] Martel D, Lauze M, Agnoux A, Fruteau de Laclos L, Daoust R, Emond M, Sirois MJ, Aubertin-Leheudre M. Comparing the effects of a home-based exercise program using a gerontechnology to a community-based group exercise program on functional capacities in older adults after a minor injury. Exp Gerontol. 2018 Jul 15;108:41-47. doi: 10.1016/j.exger.2018.03.016. Epub 2018 Mar 22. No abstract available. PMID 29577975
- [Background] Barbosa Neves B, Franz R, Judges R, Beermann C, Baecker R. Can Digital Technology Enhance Social Connectedness Among Older Adults? A Feasibility Study. J Appl Gerontol. 2019 Jan;38(1):49-72. doi: 10.1177/0733464817741369. Epub 2017 Nov 22. PMID 29166818
- [Background] Angarita-Fonseca A, Page MG, Meloto CB, Gentile EL, Leonard G, Masse-Alarie H, Tufa I, Roy JS, Stone LS, Choiniere M, Fortin M, Roy M, Sean M, Tetreault P, Rainville P, Deslauriers S, Lacasse A; Quebec Back Pain Consortium; Quebec Back Pain Consortium. The Canadian version of the National Institutes of Health minimum dataset for chronic low back pain research: reference values from the Quebec Low Back Pain Study. Pain. 2023 Feb 1;164(2):325-335. doi: 10.1097/j.pain.0000000000002703. Epub 2022 Jun 2. PMID 36638305
- See also: Fitbit news. The impact of coronavirus on Global activity, March 23, 2020 — https://blog.fitbit.com/covid-19-global-activity/?fbclid=IwAR30cP5nVULDV2oIlfYvTKcCw2v1u7uw7S84Abzn8oFBnmm7umaMtCfLdLg)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT05895630/Prot_SAP_000.pdf